CLINICAL TRIAL: NCT03529695
Title: In-home Obesity Prevention to Reach Low-income Infants Through Maternal and Social Transmission
Brief Title: In-home Obesity Prevention to Reach Low-income Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Antelope Valley Partners for Health (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Kayla de la Haye, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD092483-01 (NIH); 1R01HD092483-01 (NIH)
Record Dates: First submitted 2018-04-20; First posted 2018-05-18 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Obesity, Childhood; Obesity; Familial
Keywords: obesity; childhood obesity; maternal and child health; health disparities; prevention; low-income; social network; home environment
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomization occurs at the level of home visitors who deliver the home visitation program curriculum. Home visitors will be randomized to deliver the home visitation program curriculum with (Experimental comparator) or without (Active Comparator) the obesity prevention enhancement module. Mother-child dyads enrolled in home visitation programs, and who agree to participate in the study, will receive the intervention arm delivered by their home visitor.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard HVP Curriculum (Active Comparator): Participants will receive the standard Healthy Families America (HFA) home visitation curriculum delivered by trained home visitors. The HFA model meets the Department of Health and Human Services criteria for an "evidence-based early childhood home visiting service delivery model". HFA services begin prenatally and continue until children are 2-5yo. The curriculum focuses on strengthening parent-child relationships and family functioning, promoting positive child development, and linkage to community resources. Accredited home visitors are matched to families on cultural background and language, to provide culturally sensitive services. Home visitors receive weekly supervision, ongoing developmental training, and have limited caseloads (10-15 families) to meet their families' needs.
  Interventions: Behavioral: Standard HVP Curriculum
- Obesity Prevention (Experimental): Participants will receive the standard Healthy Families America home visitation curriculum with the obesity prevention enhancement module, delivered by trained home visitors. Families are matched to home visitors based on their ethnicity/race and language preferences. The obesity prevention program targets 4 key behaviors (physical activity, fruit and vegetable consumption, sugary beverages, fried foods) aimed at reducing obesity risks in mothers and their children. Participants will also be provided opportunities to meet in groups with other participating mothers/infants to enhance social networks that support healthy eating and physical activity.
  Interventions: Behavioral: Standard HVP Curriculum; Behavioral: Obesity Prevention

INTERVENTIONS:
Behavioral: Standard HVP Curriculum — Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
Behavioral: Obesity Prevention — Obesity prevention curriculum program targets 4 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, and decreasing fried foods) aimed at reducing obesity risk in mothers and children. The module will also include weekly activity opportunities to develop social networks that foster healthy eating and physical activity.
  Arms: Obesity Prevention

SUMMARY:
Existing obesity prevention efforts have had limited success among underserved, low-income children. This study capitalizes on the strengths of a nationwide ongoing Home Visitation Program (HVP), which serves at-risk, low-income, ethnically/racially diverse mothers and their infants, to test the effectiveness of delivering obesity prevention as part of their weekly, in-home services. The study will evaluate whether the integration of an obesity prevention enhancement module into existing HVP services, reduces the risk and incidence of obesity and associated risk factors in mothers and infants, compared to the provision of standard home visitation services. The study also focuses on the role of maternal factors (maternal diet, physical activity, food insecurity and feeding practices) and social factors (social network support) as mechanisms operating on infant outcomes.

DETAILED DESCRIPTION:
More than 40% of children enrolled in federally funded programs are overweight or obese by age 5. Unfortunately, extant obesity efforts have had a limited impact among low-income underserved children, in part because of limitations inherent to existing programs: 1) short duration and low intensity; 2) late timing of implementation, when children are already overweight or obese; 3) delivery methods limiting their accessibility and sustainability; and 4) failure to address barriers such as a lack of culturally competent services, poverty, housing instability, and access to care, which interfere with healthy lifestyle changes. To address these gaps, we have integrated simple, evidence-based nutrition and physical activity components as part of the services already delivered by our home visitation partner, Healthy Families America, with the long-term goal to deploy these efforts to Home Visitation Programs (HVPs) nationwide. Annually, over 500 publicly and privately funded HVPs provide nationwide services to more than 650,000 low-income, underserved infants and their families. The home visiting structure is not only an unparalleled model for scalable and sustainable childhood obesity prevention, but it also provides a unique opportunity to understand factors related to the intergenerational transmission of obesity in families who are most at risk.

Over the last four years, our transdisciplinary team of researchers, home visiting stakeholders, families, and community stakeholders has integrated evidence-based nutrition and physical activity components into an engaging obesity prevention curriculum delivered in English and Spanish as an enhancement module to the services of our HVP partner. Our pilot work supports the successful integration, feasibility, and preliminary efficacy of integrating obesity prevention as part of HVP services. The proposed study tests the large-scale and sustained impact of home-based obesity prevention on infant's and mothers' obesity outcomes, and studies key mechanisms of maternal and social transmission on infants' obesity risk.

Specifically, 300 low-income mothers/infants enrolled in Healthy Families America's HVP will be recruited and enrolled in the study. Based on standard HVP procedures, mothers/infants will be matched to highly trained home visitors based on their ethnicity/race and language preferences. Home visitors, in turn, will be randomly assigned to deliver the standard HVP curriculum only or the standard HVP curriculum + obesity prevention as part of their weekly home visits, for the first 12 months of HVP services. Comprehensive assessments of mothers/infants will be conducted at enrollment and after 6 and 12 months of intervention.

Aim 1 (maternal and infant outcomes). Test the direct effects of obesity prevention on infants and mothers' weight, metabolic risks, diet/energy intake, and physical activity. This will be accomplished by comparing changes in body weight, metabolic markers, and eating and activity-related behaviors between infants/mothers across study arms (HVP only vs. HVP+obesity prevention). These results will indicate whether HVP is an effective infrastructure for primary and secondary obesity prevention.

Aim 2 (maternal transmission). Test whether breastfeeding and maternal diet and activity, feeding practices, and food insecurity mediate the effect of obesity prevention on infants' outcomes. This aim will test mechanisms of maternal transmission on infants' obesity risks.

Aim 3 (social transmission). Aim 3 is two-pronged. Aim 3a tests the direct effect of HVP+obesity prevention (vs. HVP only) on the characteristics of the social and community networks that surround mothers and infants (i.e., the density, composition, and quality of health support networks). Aim 3b tests whether the characteristics of social networks mediate the effects of obesity prevention on maternal and infant outcomes. These findings will indicate if the delivery of in-home obesity prevention efforts can alter and/or activate social network mechanisms.

Secondary Aim. Conduct a real-life economic analysis (costs, cost-savings, and non-monetary benefits) of integrating obesity prevention into existing HVPs.

This proposal addresses the impetus to develop interventions targeting at-risk infants before obesity is established. Although maternal-infant interventions are much-needed, they present implementation and dissemination challenges, including limitations on compliance and retention, and limited potential for scalability and sustainability. Our proposed strategy overcomes these challenges through an innovative solution that merges evidence-based nutrition and activity components into an existing, ongoing federally-funded infrastructure. The proposed research is timely as the Institute of Medicine, the United States Department of Agriculture, and Health and Human Services (DHHS) extend their recommendations to address key factors influencing obesity risk in children from birth to 24 months of age.

ELIGIBILITY:
*Important: Mother (or caregiver) and child dyads are enrolled together. Both must meet inclusion criteria to participate.

Inclusion Criteria:

Mothers:

* Enrolled in a partnered home visitation program
* Mother or primary caregiver of 2-8 month old child
* BMI above 18.5
* Generally Healthy

Children:

* 2-8 months of age at time of enrollment
* Parent or primary caregiver receiving home visitation services

Exclusion Criteria:

Mothers:

* Any history of an eating or feeding disorder, or obesity related syndrome (such as Prader-Willi)
* Diagnosis of Schizophrenia
* Currently enrolled in a diet and weight loss program, AND either a) significant weight loss of 10+ pounds in the last 6 months, OR b) unwilling to discontinue from current diet and weight loss program.

Infants:

* Infant is clinically underweight (<5th percentile) or has a history of a feeding or eating disorder

Min Age: 2 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kayla de la Haye, PhD, Principal Investigator — University of Southern California; Sarah-Jeanne Salvy, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Development, execution, and data collection for this study is completed with a Principle Investigator at Cedars-Sinai Medical Center. Data will be shared with Dr. Salvy and her staff as appropriate. With documented permission of the IRB, a PI may develop a de-identified database, codebook, and mechanism by which data can be shared with qualified investigators. Interested Investigators will complete a request form stating the aims of their analyses, analytic plan, available resources for completing a project, timeline, and goals (i.e. manuscripts or grant applications). The PIs and their research team will review requests to determine whether the analyses constitute an innovative exploration of the data, whether the team has resources to complete the request, and whether data will be adequately protected and managed. If issues arise, the PIs and research team will negotiate a fair resolution with interested investigators and NIH staff.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed, and requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] de la Haye K, Fluke M, Laney PC, Goran M, Galama T, Chou CP, Salvy SJ. In-home obesity prevention in low-income infants through maternal and social transmission. Contemp Clin Trials. 2019 Feb;77:61-69. doi: 10.1016/j.cct.2018.12.010. Epub 2018 Dec 19. PMID 30578850

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mother-child dyads were recruited into the study. Home visitors who delivered the program in the intervention and control arms were not enrolled into the study.
Pre-assignment Details: The enrollment number represents the number of mother-infant dyads.
Groups:
- Standard HVP Curriculum- Mothers; Standard HVP Curriculum - Children: Mother and their children participants will receive the standard Healthy Families America (HFA) home visitation curriculum delivered by trained home visitors. The HFA model meets the Department of Health and Human Services criteria for an "evidence-based early childhood home visiting service delivery model". HFA services begin prenatally and continue until children are 2-5yo. The curriculum focuses on strengthening parent-child relationships and family functioning, promoting positive child development, and linkage to community resources. Accredited home visitors are matched to families on cultural background and language, to provide culturally sensitive services. Home visitors receive weekly supervision, ongoing developmental training, and have limited caseloads (10-15 families) to meet their families' needs.
  Standard HVP Curriculum: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
- Obesity Prevention - Mothers; Obesity Prevention - Children: Mother and their children participants will receive the standard Healthy Families America home visitation curriculum with the obesity prevention enhancement module, delivered by trained home visitors. Families are matched to home visitors based on their ethnicity/race and language preferences. The obesity prevention program targets 4 key behaviors (physical activity, fruit and vegetable consumption, sugary beverages, fried foods) aimed at reducing obesity risks in mothers and their children. Participants will also be provided opportunities to meet in groups with other participating mothers/infants to enhance social networks that support healthy eating and physical activity.
  Standard HVP Curriculum: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
  Obesity Prevention: Obesity prevention curriculum program targets 4 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, and decreasing fried foods) aimed at reducing obesity risk in mothers and children. The module will also include weekly activity opportunities to develop social networks that foster healthy eating and physical activity.
Period: Overall Study
Arm/Group | Standard HVP Curriculum- Mothers | Obesity Prevention - Mothers | Standard HVP Curriculum - Children | Obesity Prevention - Children
Started | 35 | 42 | 35 | 42
Completed | 20 | 22 | 20 | 22
Not Completed | 15 | 20 | 15 | 20

BASELINE CHARACTERISTICS:
Population: Baseline data obtained for 76 mother-child dyads (152 participants total)
Groups:
- Standard HVP Curriculum-Mothers; Standard HVP Curriculum-Children: Participants will receive the standard Healthy Families America (HFA) home visitation curriculum delivered by trained home visitors. The HFA model meets the Department of Health and Human Services criteria for an "evidence-based early childhood home visiting service delivery model". HFA services begin prenatally and continue until children are 2-5yo. The curriculum focuses on strengthening parent-child relationships and family functioning, promoting positive child development, and linkage to community resources. Accredited home visitors are matched to families on cultural background and language, to provide culturally sensitive services. Home visitors receive weekly supervision, ongoing developmental training, and have limited caseloads (10-15 families) to meet their families' needs.
  Standard HVP Curriculum: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
- Obesity Prevention-Mothers; Obesity Prevention-Children: Participants will receive the standard Healthy Families America home visitation curriculum with the obesity prevention enhancement module, delivered by trained home visitors. Families are matched to home visitors based on their ethnicity/race and language preferences. The obesity prevention program targets 4 key behaviors (physical activity, fruit and vegetable consumption, sugary beverages, fried foods) aimed at reducing obesity risks in mothers and their children. Participants will also be provided opportunities to meet in groups with other participating mothers/infants to enhance social networks that support healthy eating and physical activity.
  Standard HVP Curriculum: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
  Obesity Prevention: Obesity prevention curriculum program targets 4 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, and decreasing fried foods) aimed at reducing obesity risk in mothers and children. The module will also include weekly activity opportunities to develop social networks that foster healthy eating and physical activity.
- Total: Total of all reporting groups
Arm/Group | Standard HVP Curriculum-Mothers | Obesity Prevention-Mothers | Standard HVP Curriculum-Children | Obesity Prevention-Children | Total
Number analyzed (Participants) | 34 | 42 | 34 | 42 | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (6.4) | 29.7 (7.3) | 0.875 (0.625) | 0.825 (0.767) | 15.05 (3.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 42 | 17 | 24 | 117
  Male | 0 | 0 | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 27 | 22 | 28 | 102
  Not Hispanic or Latino | 9 | 13 | 11 | 11 | 44
  Unknown or Not Reported | 0 | 2 | 1 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 1 | 4
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 7 | 6 | 26
  White | 15 | 19 | 16 | 16 | 66
  More than one race | 1 | 3 | 4 | 7 | 15
  Unknown or Not Reported | 9 | 12 | 6 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mother BMI
Description: Body mass index (BMI) at each assessment
Time Frame: Baseline, 6 months, 12 months
Population: Some participants did not compete all study assessments.
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Obesity Prevention: Participants will receive the standard Healthy Families America home visitation curriculum with the obesity prevention enhancement module, delivered by trained home visitors. Families are matched to home visitors based on their ethnicity/race and language preferences. The obesity prevention program targets 4 key behaviors (physical activity, fruit and vegetable consumption, sugary beverages, fried foods) aimed at reducing obesity risks in mothers and their children. Participants will also be provided opportunities to meet in groups with other participating mothers/infants to enhance social networks that support healthy eating and physical activity.
  Standard HVP Curriculum: The content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
  Obesity Prevention: Obesity prevention curriculum program targets 4 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, and decreasing fried foods) aimed at reducing obesity risk in mothers and children. The module will also include weekly activity opportunities to develop social networks that foster healthy eating and physical activity.
Arm/Group | Standard HVP Curriculum | Obesity Prevention
Number analyzed (Participants) | 31 | 40
kg/m^2
  Baseline | 30.6 (8.1) | 34.2 (9.5)
  6 Month: number analyzed (Participants) | 18 | 20
  6 Month | 34 (8.7) | 34.3 (9.8)
  12 Month: number analyzed (Participants) | 8 | 13
  12 Month | 32 (9.6) | 35.4 (10)

2. Primary Outcome: Infant Weight
Description: weight in pounds
Time Frame: Baseline, 6 months, 12 months
Population: Missing data
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Standard HVP Curriculum | Obesity Prevention
Number analyzed (Participants) | 34 | 42
pounds
  Baseline: number analyzed (Participants) | 30 | 35
  Baseline | 20.0 (5.7) | 19.3 (6.5)
  6 Month: number analyzed (Participants) | 19 | 18
  6 Month | 24.2 (5.6) | 22.1 (3.3)
  12 Months: number analyzed (Participants) | 18 | 17
  12 Months | 30.3 (10.1) | 28.9 (5.8)

3. Secondary Outcome: Fruit Intake Frequency
Description: Assessed using modified food frequency measures from the National Health and Nutrition Examination Survey (NHANES).
Time Frame: Baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Standard HVP Curriculum - Mothers; Standard HVP Curriculum - Children: Participants will receive the standard Healthy Families America (HFA) home visitation curriculum delivered by trained home visitors. The HFA model meets the Department of Health and Human Services criteria for an "evidence-based early childhood home visiting service delivery model". HFA services begin prenatally and continue until children are 2-5yo. The curriculum focuses on strengthening parent-child relationships and family functioning, promoting positive child development, and linkage to community resources. Accredited home visitors are matched to families on cultural background and language, to provide culturally sensitive services. Home visitors receive weekly supervision, ongoing developmental training, and have limited caseloads (10-15 families) to meet their families' needs.
  Standard HVP Curriculum: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
- Obesity Prevention - Mothers; Obesity Prevention - Children: Participants will receive the standard Healthy Families America home visitation curriculum with the obesity prevention enhancement module, delivered by trained home visitors. Families are matched to home visitors based on their ethnicity/race and language preferences. The obesity prevention program targets 4 key behaviors (physical activity, fruit and vegetable consumption, sugary beverages, fried foods) aimed at reducing obesity risks in mothers and their children. Participants will also be provided opportunities to meet in groups with other participating mothers/infants to enhance social networks that support healthy eating and physical activity.
  Standard HVP Curriculum: The content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
  Obesity Prevention: Obesity prevention curriculum program targets 4 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, and decreasing fried foods) aimed at reducing obesity risk in mothers and children. The module will also include weekly activity opportunities to develop social networks that foster healthy eating and physical activity.
Arm/Group | Standard HVP Curriculum - Mothers | Obesity Prevention - Mothers | Standard HVP Curriculum - Children | Obesity Prevention - Children
Number analyzed (Participants) | 34 | 42 | 34 | 42
Participants
  Baseline: Less than once a week | 7 | 3 | 13 | 21
  Baseline: 1 to 6 times a week | 11 | 17 | 10 | 6
  Baseline: 1 or more times a day | 16 | 22 | 11 | 15
  Baseline: Missing | 0 | 0 | 0 | 0
  6 months: Less than once a week | 4 | 5 | 1 | 2
  6 months: 1 to 6 times a week | 12 | 13 | 6 | 8
  6 months: 1 or more times a day | 8 | 7 | 17 | 13
  6 months: Missing | 10 | 17 | 10 | 19
  12 months: Less than once a week | 2 | 3 | 0 | 0
  12 months: 1 to 6 times a week | 11 | 9 | 10 | 6
  12 months: 1 or more times a day | 7 | 10 | 10 | 16
  12 months: Missing | 14 | 20 | 14 | 20

4. Secondary Outcome: Vegetable Intake Frequency
Description: Assessed using modified food and activity frequency measures from the National Health and Nutrition Examination Survey (NHANES)
Time Frame: Baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard HVP Curriculum - Mothers | Obesity Prevention - Mothers | Standard HVP Curriculum - Children | Obesity Prevention - Children
Number analyzed (Participants) | 34 | 42 | 34 | 42
Participants
  Baseline: Less than once a week | 7 | 4 | 13 | 21
  Baseline: 1 to 6 times a week | 16 | 15 | 10 | 6
  Baseline: 1 or more times a day | 11 | 23 | 11 | 15
  Baseline: Missing | 0 | 0 | 0 | 0
  6 months: Less than once a week | 4 | 3 | 2 | 1
  6 months: 1 to 6 times a week | 12 | 11 | 8 | 10
  6 months: 1 or more times a day | 8 | 10 | 14 | 14
  6 months: Missing | 10 | 18 | 10 | 17
  12 months: Less than once a week | 3 | 3 | 3 | 0
  12 months: 1 to 6 times a week | 11 | 10 | 7 | 9
  12 months: 1 or more times a day | 6 | 9 | 10 | 13
  12 months: Missing | 14 | 20 | 14 | 20

5. Secondary Outcome: Fried Food Intake Frequency
Description: as for outcome 4
Time Frame: Baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard HVP Curriculum - Mothers | Obesity Prevention - Mothers | Standard HVP Curriculum - Children | Obesity Prevention - Children
Number analyzed (Participants) | 34 | 42 | 34 | 42
Participants
  Baseline: Less than once a week | 16 | 19 | 27 | 36
  Baseline: 1 to 6 times a week | 12 | 17 | 6 | 3
  Baseline: 1 or more times a day | 6 | 5 | 1 | 3
  Baseline: Missing | 0 | 1 | 0 | 0
  6 months: Less than once a week | 10 | 9 | 19 | 21
  6 months: 1 to 6 times a week | 10 | 11 | 5 | 4
  6 months: 1 or more times a day | 4 | 5 | 0 | 0
  6 months: Missing | 10 | 17 | 10 | 17
  12 months: Less than once a week | 10 | 14 | 13 | 17
  12 months: 1 to 6 times a week | 9 | 7 | 7 | 4
  12 months: 1 or more times a day | 1 | 1 | 0 | 1
  12 months: Missing | 14 | 20 | 14 | 20

6. Secondary Outcome: Soda Intake Frequency
Description: as for outcome 4
Time Frame: Baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard HVP Curriculum - Mothers | Obesity Prevention - Mothers | Standard HVP Curriculum - Children | Obesity Prevention - Children
Number analyzed (Participants) | 34 | 42 | 34 | 42
Participants
  Baseline: Less than once a week | 20 | 21 | 31 | 42
  Baseline: 1 to 6 times a week | 9 | 16 | 2 | 0
  Baseline: 1 or more times a day | 5 | 5 | 0 | 0
  Baseline: Missing | 0 | 0 | 1 | 0
  6 months: Less than once a week | 15 | 15 | 22 | 24
  6 months: 1 to 6 times a week | 7 | 8 | 2 | 1
  6 months: 1 or more times a day | 2 | 2 | 0 | 0
  6 months: Missing | 10 | 17 | 10 | 17
  12 months: Less than once a week | 12 | 18 | 19 | 21
  12 months: 1 to 6 times a week | 4 | 2 | 0 | 1
  12 months: 1 or more times a day | 3 | 2 | 0 | 0
  12 months: Missing | 15 | 20 | 15 | 20

7. Secondary Outcome: Fruit Juice Intake Frequency
Description: as for outcome 4
Time Frame: Baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard HVP Curriculum - Mothers | Obesity Prevention - Mothers | Standard HVP Curriculum - Children | Obesity Prevention - Children
Number analyzed (Participants) | 34 | 42 | 34 | 42
Participants
  Baseline: Less than once a week | 18 | 12 | 24 | 32
  Baseline: 1 to 6 times a week | 10 | 22 | 7 | 5
  Baseline: 1 or more times a day | 6 | 8 | 3 | 5
  Baseline: Missing | 0 | 0 | 0 | 0
  6 months: Less than once a week | 10 | 12 | 11 | 15
  6 months: 1 to 6 times a week | 8 | 10 | 9 | 6
  6 months: 1 or more times a day | 6 | 3 | 4 | 4
  6 months: Missing | 10 | 17 | 10 | 17
  12 months: Less than once a week | 15 | 8 | 11 | 7
  12 months: 1 to 6 times a week | 3 | 9 | 6 | 10
  12 months: 1 or more times a day | 2 | 5 | 3 | 5
  12 months: Missing | 14 | 20 | 14 | 20

8. Secondary Outcome: Mother Movement Frequency
Description: Assessed using modified activity frequency measures from the National Health and Nutrition Examination Survey (NHANES)
Time Frame: Baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard HVP Curriculum | Obesity Prevention
Number analyzed (Participants) | 34 | 42
Participants
  Baseline: 2 times a day or less | 8 | 8
  Baseline: 3 to 7 times a day | 13 | 12
  Baseline: 8 or more times a day | 10 | 17
  Baseline: Missing | 3 | 5
  6 months: 2 times a day or less | 4 | 4
  6 months: 3 to 7 times a day | 10 | 9
  6 months: 8 or more times a day | 6 | 9
  6 months: Missing | 14 | 20
  12 months: 2 times a day or less | 6 | 4
  12 months: 3 to 7 times a day | 8 | 10
  12 months: 8 or more times a day | 6 | 7
  12 months: Missing | 14 | 21

9. Secondary Outcome: Frequency of Infant Supervised Active Movement (Activity)
Description: as for outcome 4
Time Frame: Baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard HVP Curriculum | Obesity Prevention
Number analyzed (Participants) | 34 | 42
Participants
  Baseline: Less than once a week | 1 | 5
  Baseline: 1 to 6 times a week | 6 | 11
  Baseline: 1 or 2 times a day | 5 | 9
  Baseline: 3 or more times a day | 19 | 13
  Baseline: Missing | 3 | 4
  6 months: Less than once a week | 0 | 1
  6 months: 1 to 6 times a week | 2 | 8
  6 months: 1 or 2 times a day | 5 | 3
  6 months: 3 or more times a day | 13 | 10
  6 months: Missing | 14 | 20
  12 months: Less than once a week | 1 | 2
  12 months: 1 to 6 times a week | 5 | 3
  12 months: 1 or 2 times a day | 10 | 14
  12 months: 3 or more times a day | 4 | 3
  12 months: Missing | 14 | 20

10. Other Pre Specified Outcome: Maternal Food Security
Description: The U.S. Adult Food Security Survey Module will be used to evaluate hunger and food sufficiency to meet the basic needs of families.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Maternal Social Isolation
Description: Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) short form scale for social isolation.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Maternal Instrumental Support
Description: Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) short form scale for instrumental support.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Maternal Emotional Support
Description: Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) short form scale for emotional support.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Social Network Health Norms
Description: The characteristics of the social actors (people) and relationships that surround mothers will be assessed using egocentric social network methods and social network analysis (SNA) to compute the health behavior and weight norms.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Social Network Support
Description: The characteristics of the social actors (people, organizations) and relationships that surround mothers will be assessed using egocentric social network methods and social network analysis (SNA) to compute the density of relationships that provide health-related social support.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Household Activity Environment
Description: Household environment assessing availability, accessibility, and visibility of activity items will be assessed using a modified Home Food Assessment (HFA) and Home - Inventory Describing Eating and Activity Development (H-IDEA), relating to the target activity behaviors.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Household Food Environment
Description: Household environment assessing availability, accessibility, and visibility of food items will be assessed using a modified Home Food Assessment (HFA) and Home - Inventory Describing Eating and Activity Development (H-IDEA), relating to the target eating behaviors.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Habit Strength of Maternal Eating, Activity, and Feeding Behaviors
Description: Habit strength will be assessed using the Self-Reported Habit Index (SRHI) specific to target eating and activity behaviors.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Demographic History
Description: Self-reported demographic history (gender, age, race, household income, etc) will be collected. Acculturation is measured using the Demographic Index of Cultural Exposure (DICE).
Time Frame: Baseline
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Medical History
Description: Self-reported medical history (prescription medications, child and parent/caregiver illnesses, etc.) will be collected
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Depression
Description: The Edinburgh Postnatal Depression Scale (EPDS) will be used to determine maternal depression. Each of the 10 items has 4 optional responses with a set coding frame. Scores are summed and can range from 0 to 30. Values over 11 are indicative of risk for postnatal depression.
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Mother's Blood Pressure
Description: Blood pressure will be collected prior to all blood draws
Time Frame: Baseline, 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 years
Description: Adverse event information was systematically collected and reported to IRB.
Groups:
- Standard HVP Curriculum-Children: Child participants will receive the standard Healthy Families America (HFA) home visitation curriculum delivered by trained home visitors. The HFA model meets the Department of Health and Human Services criteria for an "evidence-based early childhood home visiting service delivery model". HFA services begin prenatally and continue until children are 2-5yo. The curriculum focuses on strengthening parent-child relationships and family functioning, promoting positive child development, and linkage to community resources. Accredited home visitors are matched to families on cultural background and language, to provide culturally sensitive services. Home visitors receive weekly supervision, ongoing developmental training, and have limited caseloads (10-15 families) to meet their families' needs.
  Standard HVP Curriculum: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
- Obesity Prevention-Children: Child participants will receive the standard Healthy Families America home visitation curriculum with the obesity prevention enhancement module, delivered by trained home visitors. Families are matched to home visitors based on their ethnicity/race and language preferences. The obesity prevention program targets 4 key behaviors (physical activity, fruit and vegetable consumption, sugary beverages, fried foods) aimed at reducing obesity risks in mothers and their children. Participants will also be provided opportunities to meet in groups with other participating mothers/infants to enhance social networks that support healthy eating and physical activity.
  Standard HVP Curriculum: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on strengthening children's cognitive skills, early literacy skills, social/emotional and physical development.
  Obesity Prevention: Obesity prevention curriculum program targets 4 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, and decreasing fried foods) aimed at reducing obesity risk in mothers and children. The module will also include weekly activity opportunities to develop social networks that foster healthy eating and physical activity.
Arm/Group | Standard HVP Curriculum-Mothers | Obesity Prevention-Mothers | Standard HVP Curriculum-Children | Obesity Prevention-Children
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/42 | 0/35 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/42 | 0/35 | 0/42
Other Adverse Events (participants affected / at risk) | 2/35 | 1/42 | 2/35 | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard HVP Curriculum-Mothers (N=35) | Obesity Prevention-Mothers (N=42) | Standard HVP Curriculum-Children (N=35) | Obesity Prevention-Children (N=42)
Breach of Confidentiality (Social circumstances) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Data Deletion (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Survey data mistakenly deleted from server

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT03529695/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT03529695/ICF_001.pdf